CLINICAL TRIAL: NCT04804553
Title: A Phase 3, Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Apremilast in Children From 5 to Less Than 18 Years of Age With Active Juvenile Psoriatic Arthritis (PEAPOD)
Brief Title: Apremilast Pediatric Study in Children With Active Juvenile Psoriatic Arthritis
Acronym: PEAPOD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20190529
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Active Juvenile Psoriatic Arthritis
Keywords: Apremilast; Otezla®; Juvenile psoriatic arthritis; Inflammatory disorders
MeSH Terms: conditions — Arthritis, Juvenile | interventions — apremilast

STUDY DESIGN:
Intervention Model Description: The participants will be randomized to receive apremilast or placebo in the double-blind 16 week treatment phase. Then, the participants will all receive apremilast for a further 36 weeks in the active treatment phase. The participants not continuing to receive apremilast through the Post-Trial Access Program or Open-label Extension study will then complete the 30 days safety follow-up period after the last dose of apremilast in the active treatment phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Apremilast (Experimental): Participants will receive apremilast in the double-blind 16 week treatment phase. Then the participants will continue to receive apremilast in the active 36 weeks treatment phase.
  Interventions: Drug: Apremilast
- Placebo to Apremilast (Placebo Comparator): Participants will receive the matching placebo in the double-blind 16 week treatment phase. Then the participants will receive apremilast in the active 36 weeks treatment phase.
  Interventions: Drug: Apremilast; Drug: Placebo

INTERVENTIONS:
Drug: Apremilast — Participants will receive apremilast orally.
  Other Names: Otezla®
Drug: Placebo — Participants will receive the matching placebo orally.
  Arms: Placebo to Apremilast

SUMMARY:
The study will aim to estimate the efficacy of apremilast compared with placebo in the treatment of juvenile psoriatic arthritis (JPsA) in pediatric participants 5 to less than 18 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female participants 5 to < 18 years of age at the time of randomization.
* Participant must have a confirmed diagnosis of juvenile psoriatic arthritis (JPsA) according to the International League of Associations for Rheumatology (ILAR) Edmonton Revision (Petty, 2001) classification criteria of at least 6 months duration:

  * Arthritis and psoriasis, OR
  * Arthritis with at least 2 of the following:
  * Dactylitis
  * Nail pitting or onycholysis
  * Psoriasis in a first-degree relative
* Active disease: at least 3 active joints.
* Inadequate response (at least 2 months) or intolerance to ≥ 1 disease-modifying anti-rheumatic drugs (DMARD), (which may include methotrexate [MTX] or biologic agents).

Exclusion Criteria:

* Exclusions per ILAR Edmonton Revision (Edmonton, 2001) criteria for JPsA include:

  * Arthritis in an HLA-B27-positive male with arthritis onset after 6 years of age
  * Ankylosing spondylitis, sacroiliitis with inflammatory bowel disease, Reiter's syndrome, acute anterior uveitis, or a history of one of these disorders in a first-degree relative
  * History of IgM rheumatoid factor on at least 2 occasions at least 3 months apart
  * Presence of systemic juvenile idiopathic arthritis (JIA).
* Rheumatic autoimmune disease other than psoriatic arthritis (PsA), including, but not limited to: systemic lupus erythematosus, mixed connective tissue disease, scleroderma, polymyositis, or fibromyalgia.
* Prior history of or current inflammatory joint disease other than PsA (eg, gout, reactive arthritis, rheumatoid arthritis, ankylosing spondylitis, Lyme disease).

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2028-03-21 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Achieve American College of Rheumatology Pediatric (ACR) Pedi 30 Response at Week 16 | Baseline to Week 16
  The ACR Pedi 30 is defined as a minimum of 30 percent improvement from baseline in a minimum of 3 out of 6 components, with no more than 1 component worsening by >30 percent.
  The ACR Pedi consists of 6 core criteria:
  1. physician global assessment (PGA) of disease activity (visual analog scale [VAS]) where 0 represents no disease activity and 100 represents the most disease activity
  2. assessment of overall well-being (VAS) where 0 represents very well and 100 represents very poor for overall well-being
  3. functional ability (assessed using the Childhood Health Assessment Questionnaire [CHAQ]);
  4. number of joints with active arthritis (defined as joints with swelling not caused by deformity or joints, in the absence of swelling, with limitation of passive motion accompanied by pain, tenderness, or both)
  5. number of joints with limited range of motion
  6. laboratory marker of inflammation (C-reactive protein [CRP]).

SECONDARY OUTCOMES:
Change from Baseline in Participants Assessment of Pain at Week 16 | Baseline to Week 16
  The participants assessment of pain will be assessed using a visual analogue scale (VAS). Participants will be asked to place a vertical line on a 100-mm VAS where the left-hand boundary represents "no pain" and the right-hand boundary represents "worst possible pain".
Number of Participants who Achieve ACR Pedi 20, ACR Pedi 50, ACR Pedi 70 and ACR Pedi 90 Response at Week 16 | Baseline to Week 16
  The ACR Pedi 20, 50, 70 and 90 is defined as a minimum of either 20 percent, 50 percent. 70 percent or 90 percent improvement respectively from baseline in a minimum of 3 out of 6 components, with no more than 1 component worsening by >20 percent, >50 percent, >70 percent or >90 percent respectively.
  The ACR Pedi consists of 6 core criteria:
  1. PGA of disease activity (VAS) where 0 represents no disease activity and 100 represents the most disease activity
  2. assessment of overall well-being (VAS) where 0 represents very well and 100 represents very poor for overall well-being
  3. functional ability (assessed using the CHAQ)
  4. number of joints with active arthritis (defined as joints with swelling not caused by deformity or joints, in the absence of swelling, with limitation of passive motion accompanied by pain, tenderness, or both) 5. number of joints with limited range of motion
  6. laboratory marker of inflammation (CRP).
Change from Baseline in the Physician Global Assessment (PGA) of Disease Activity at Week 16 | Baseline to Week 16
  PGA of disease activity is assessed using a visual analog scale (VAS), where 0 represents no disease activity and 100 represents the most disease activity.
Change from Baseline in the Assessment of Overall Well-being at Week 16 | Baseline to Week 16
  Assessment of overall well-being is assessed using a visual analog scale (VAS), where 0 represents very well and 100 represents very poor for overall well-being. This assessment can be completed by either the participant or the parent/caregiver.
Change from Baseline in the Number of Joints with Active Arthritis at Week 16 | Baseline to Week 16
  Active arthritis is defined as joints with swelling not caused by deformity of joints, in the absence of swelling, with limitation of passive motion accompanied by pain, tenderness, or both.
Change from Baseline in the Number of Joints with Limited Range of Motion at Week 16 | Baseline to Week 16
Change from Baseline in the Laboratory Marker of Inflammation (C-reactive Protein) at Week 16 | Baseline to Week 16
Change from Baseline in Childhood Health Assessment Questionnaire (CHAQ) at Week 16 | Baseline to Week 16
  The CHAQ will be used to assess physical ability and functional status of participants as well as their quality of life.
  The CHAQ consists of 20 items concerning difficulty in performing the following 8 activities of daily living: dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping, and activities. Subjects will choose from 4 responses ranging from 0 (without any difficulty) to 3 (unable to do). A lower score indicates a better outcome. The subject's/parent's/caregiver's assessment of arthritis-related pain will also be assessed on a VAS that is part of the CHAQ.
Change from Baseline in Juvenile Arthritis Disease Activity Score (JADAS) at Week 16 | Baseline to Week 16
  JADAS is a composite score of participant well-being visual analog scale (VAS) score, physician global assessment (PGA) VAS score, active joint count, and laboratory marker of inflammation (C-reactive protein [CRP]).
  There are 4 components of the JADAS:
  1. Active joint count (71 joints)
  2. PGA (0 to 100) measured on a VAS
  3. Patient/parent global assessment of well-being (0 to 100) measured on a VAS
  4. CRP (normalized to a 0 to 10 scale)
  The active joint count is taken from 71 joints: Temporomandibular joints, cervical spine, glenohumeral joints, acromioclavicular joints, sternoclavicular joints, elbows, wrists, metacarpophalangeal joints, interphalangeal joints, proximal interphalangeal joints, distal interphalangeal joints, hips, subtalar joints, midfoot joints, knees and ankles .
  The total score is calculated by adding all 4 components of the JADAS. The score for the JADAS ranges from 0 to 101 where a lower score indicates a better outcome.
Number of Participants who Experience Psoriatic Arthritis (PsA) Flares at Week 16 | Baseline to Week 16
  PsA flares are defined as more than or equal to 30 percent worsening in at least 3 of 6 American College of Rheumatology Pediatric (ACR Pedi) core set variables with a more than or equal to 30 percent improvement in not more than 1 of 6 ACR Pedi core set variables.
Psoriasis Area Severity Index (PASI)-75 Response at Week 16 for Participants With a Baseline Psoriasis Body Surface Area (BSA) ≥ 3 percent | Baseline to Week 16
  PASI scores range from 0 to 72, with higher scores reflecting greater disease severity.
  The PASI score is determined only for subjects whose BSA involved by psoriasis is
  ≥3 percent. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on the 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90 percent < 100 percent involvement). The sum of scores for erythema, thickness, and scaling is multiplied by the degree of involvement for each anatomic region, and then multiplied by a constant corresponding to the region's percentage of BSA. The resultant values for each anatomic region are then summed to yield the PASI score.
Number of Participants who Experience One or More Treatment-Emergent Adverse Events (TEAEs) | Up to Week 56
Number of Participants With Suicidal Ideation or Behaviour Assessed Via the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to Week 56
  The C-SSRS is an assessment tool that evaluates suicidal ideation and behavior. Number of participants with suicidal ideation or behavior is defined as the number of participants who answer "yes" at any time during the study (up to end of safety follow-up, Week 56) to one of the 10 categories:
  Category 1: Wish to be dead Category 2: Non-specific active suicidal thoughts Category 3: Active suicidal ideation with any methods (not plan) without intent to act Category 4: Active suicidal ideation with some intent to act, without specific plan Category 5: Active suicidal ideation with specific plan and intent Category 6: Preparatory acts or behavior Category 7: Aborted attempt Category 8: Interrupted attempt Category 9: Actual attempt (non-fatal) Category 10: Completed suicide
Change from Baseline in Tanner Staging at Week 52 | Baseline to Week 52
  Tanner Staging of sexual development assessment will be used to assess sexual maturity. Tanner Staging assessment consists of 3 domains (pubic hair, breast development, and other changes) for girls and 4 domains (pubic hair, penis development, testes development, and other changes) for boys. Stages range from 1-5, with 1 indicating preadolescent and 5 adult.
Change from Baseline in Body Weight at Week 56 | Baseline to Week 56
Change from Baseline in Height at Week 56 | Baseline to Week 56
Change from Baseline in Body Mass Index (BMI) at Week 56 | Baseline to Week 56
Plasma Concentrations of Apremilast | Week 2: 0-5 hours post dose; Week 8: 2 hours post dose; Week 16: 4 hours post-dose; Week 28: pre dose; Week 40: pre dose; Week 52: pre dose
Taste and Acceptability of Apremilast | Baseline and Week 2
  Taste and acceptability will be assessed using a questionnaire with a 7-point faces Likert Scale, with 1 ranging from "super bad" to 7 "super good" and questions to determine whether the participants are able to take the treatment medication.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (45):
- Landeskrankenhaus Bregenz, Bregenz, Austria
- Belgium (3):
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Regional de la Citadelle, Liège
  - Ziekenhuis Netwerk Antwerpen Jan Palfijn, Merksem
- France (2):
  - Hospices Civils de Lyon Hopital Femme Mere Enfant, Bron
  - Hopital Jeanne de Flandre, Lille
- Germany (4):
  - Charite - Universitaetsmedizin Berlin, Campus Virchow, Berlin
  - Universitaetsklinikum Dresden, Dresden
  - An der Schoen Klinik Hamburg Eilbek, Hamburg
  - Asklepios Kinderklinik Sankt Augustin GmbH, Sankt Augustin
- Greece (3):
  - Agia Sofia Children Hospital, Athens
  - Attikon University General Hospital, Athens
  - General Hospital of Thessaloniki Ippokrateio, Thessaloniki
- Italy (4):
  - Ospedale Santissima Annunziata, Chieti
  - IRCCS Istituto Giannina Gaslini, Genova
  - Azienda Socio Sanitaria Territoriale Centro Specialistico Ortopedico Traumatologico Gaetano Pini, Milan
  - IRCCS Ospedale Pediatrico Bambino Gesu, Roma
- Viesoji istaiga Vilniaus universiteto ligonine Santaros klinikos, Vaiku ligonine, Vilnius, Lithuania
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Poland (3):
  - Wojewodzki Specjalistyczny Szpital Dzieciecy im sw Ludwika w Krakowie, Krakow
  - SPZOZ Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi, Lodz
  - Narodowy Instytut Geriatrii Reumatologii i Rehabilitacji im prof dr hab med Eleonory Reicher, Warsaw
- Portugal (5):
  - Unidade Local de Saude de Lisboa Ocidental, EPE - Hospital Egas Moniz, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
  - Unidade Local de Saude do Alto Minho EPE - Hospital do Conde de Bertiandos, Ponte de Lima
  - Unidade Local de Saude de Sao Joao, EPE - Hospital de Sao Joao, Porto
  - Unidade Local de Saude de Gaia-Espinho, EPE, Vila Nova de Gaia
- Romania (2):
  - Spitalul Clinic de Urgenta pentru Copii Cluj, Cluj-Napoca
  - Spitalul Clinic de Urgenta pentru Copii Louis Turcanu Timisoara, Timișoara
- South Africa (2):
  - Panorama Medical Centre, Panorama, Western Cape
  - Groote Schuur Hospital, Cape Town
- Spain (6):
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Canary Islands
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Catalonia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
- Turkey (Türkiye) (4):
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Umraniye Egitim ve Arastirma Hastanesi, Istanbul
- United Kingdom (4):
  - Birmingham Childrens Hospital, Birmingham
  - Alder Hey Childrens Hospital, Liverpool
  - Nottingham Childrens Hospital, Nottingham
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com